CLINICAL TRIAL: NCT07344272
Title: The Effects of Proprioceptive Neuromuscular Facilitation on Shoulder Girdle Function and Quality of Life in Individuals With Scapular Winging
Brief Title: The Effects of Proprioceptive Neuromuscular Facilitation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Bayar University (Other)
Responsible Party: Principal Investigator, Erhan Seçer, Lecturer, PT., PhD., Celal Bayar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBU-FTR-ES-O7
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Scapular Winging
Keywords: Functional status; Neuromuscular effect; Proprioceptive neuromuscular facilitation; Quality of life; Scapula
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: This study will be conducted as a randomized controlled trial. Participants will be randomly assigned to two groups: the intervention group (proprioceptive neuromuscular facilitation intervention) and the control group (no intervention).
Who Masked: Participant, Outcomes Assessor
Masking Description: The intervention group will receive proprioceptive neuromuscular facilitation and outcome measures will be assessed by an investigator who was blinded to the group allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proprioceptive Neuromuscular Facilitation Group (Active Comparator): The Proprioceptive Neuromuscular Facilitation Group will receive proprioceptive neuromuscular facilitation for a duration of 5 weeks, scheduled three times per week, with a session length of approximately 20-30 minutes.
  Interventions: Other: Proprioceptive neuromuscular facilitation
- Control Group (No Intervention): The Control Group will receive no intervention.

INTERVENTIONS:
Other: Proprioceptive neuromuscular facilitation — The Proprioceptive Neuromuscular Facilitation Group will receive proprioceptive neuromuscular facilitation for a duration of 5 weeks, scheduled three times per week, with a session length of approximately 20-30 minutes.
  Arms: Proprioceptive Neuromuscular Facilitation Group

SUMMARY:
This study aims to investigate the effects of proprioceptive neuromuscular facilitation (PNF) on shoulder girdle function and quality of life in individuals with scapular winging.

DETAILED DESCRIPTION:
Scapular stability on the thorax is fundamental for maintaining proper upper extremity function. The loss of this stability manifests clinically as scapular winging, a pathological condition characterized by the prominent protrusion of the medial (vertebral) border and/or the inferior angle of the scapula away from the thorax.

PNF can target the underlying impairment of scapular dysfunction by activating the muscle synergies required for scapulothoracic stability more powerfully and coordinately through resisted diagonal movements.

Therefore, the implementation and testing of PNF protocols are of critical importance, as this method can enhance functional strength and coordination, contributing to better clinical outcomes and improved quality of life in individuals with scapular winging.

Therefore, this study aims to investigate the effects of PNF on shoulder girdle function and quality of life in individuals with scapular winging.

In this study, designed as a randomized controlled trial, one group will receive PNF in scapular diagonals for approximately 20-30 minutes, three days a week, for a total of five weeks, to ensure scapular positioning and increase the tone of the surrounding muscles.

The control group will receive no intervention during this period.

Before (pre-test) and after (post-test) the study, participants in both groups will be evaluated using the Scapular Isometric Pinch Test for scapular muscle endurance; the Lateral Scapular Slide Test for scapular position; the Rounded Shoulder Posture Assessment for shoulder posture; the Disabilities of the Arm, Shoulder, and Hand Questionnaire for upper extremity functional level; and the Short Form-36 for quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study.
* Presenting with bilateral scapular winging (Scapular winging will be evaluated by measuring the distance between the inferior angle of the scapula and the thoracic wall using a scapulometer; a distance of ≥2 cm is considered as winging).

Exclusion Criteria:

* Presence of long thoracic nerve palsy.
* Having undergone shoulder surgery within the last 12 months or having an acute shoulder injury (e.g., rotator cuff tear, dislocation, labral pathology, etc.).
* Presence of scapulothoracic bursitis, fractures, tumors, or structural deformities in the scapular/thoracic region.
* Having received regular scapular or shoulder rehabilitation within the last 6 months.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-03-08 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Biodex System 3 Pro | one week
  Isokinetic strength measurement of the shoulder girdle muscles will be performed using a Biodex System 3 Pro isokinetic dynamometer. The measurements will be conducted in a diagonal plane specifically determined to align with scapular patterns, utilizing a concentric-concentric mode at two different angular velocities: 60°/s and 180°/s. For each test, participants will perform three trial sets; the peak torque values obtained from each set will be normalized to body weight (Nm/kg) and averaged for statistical analysis. During the test protocol, participants will be securely positioned using stabilization straps to ensure arm and trunk stability. Prior to the measurements, a device orientation and warm-up session (e.g., three practice/familiarization sets) will be conducted, followed by the actual data collection.

SECONDARY OUTCOMES:
Scapular Isometric Pinch Test | one week
  The scapular stabilizer muscles' endurance will be evaluated using the Scapular Isometric Pinch Test. During the test, participants will be asked to maintain the scapula in a bilateral retraction position and will be verbally encouraged to sustain the position for as long as they can maintain a maximal isometric contraction. The endurance time will be recorded in seconds.
The Lateral Scapular Slide Test | one week
  The Lateral Scapular Slide Test will be used to evaluate scapular dyskinesis. During the test, the participant will be positioned with their back to the researcher. The assessment will be performed bilaterally in three different upper extremity positions: i) 0° of abduction with the arms in a neutral position, (ii) 45° of abduction with the hands placed on the hips and the thumbs pointing posteriorly, and (iii) 90° of abduction with the shoulders parallel to the floor and the arms held in maximum internal rotation. In all three positions, the scapular position will be determined by measuring the distance between the inferior angle of the scapula and the spinous processes of the thoracic vertebrae.
Disabilities of the Arm, Shoulder, and Hand Questionnaire | one week
  The functional status of the upper extremity will be evaluated using the Disabilities of the Arm, Shoulder, and Hand Questionnaire. The Disabilities of the Arm, Shoulder, and Hand Questionnaireis a 30-item self-report scale that measures activities of daily living, symptom severity, and social/role functioning related to the upper extremity. Participants rate each item on a scale from 1 (no difficulty/no symptom) to 5 (unable to do/severe symptoms). The total score is transformed into a 0-100 range based on the item averages; higher scores indicate greater functional impairment.
Short Form-36 | one week
  Quality of life will be evaluated using the Short Form-36. The Short Form-36 assesses eight distinct health domains categorized under two main component summaries: Physical Functioning, Role Limitations due to Physical Problems, Bodily Pain, General Health Perceptions, Vitality, Social Functioning, Role Limitations due to Emotional Problems, and Mental Health. The scale scores range from 0 (worst health status) to 100 (best health status), with higher scores indicating a better quality of life.

IPD SHARING:
Plan to Share IPD: No